CLINICAL TRIAL: NCT06708416
Title: A Phase IIa, Randomized, Double-blind, Placebo Controlled, Parallel Group, Multi-center Trial to Evaluate the Efficacy and Safety of ONO-1110 in Patients With Postherpetic Neuralgia
Brief Title: A Study of ONO-1110 in Patients With Postherpetic Neuralgia
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Ono Pharmaceutical Co. Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ONO-1110-04; jRCT2031240504 (Registry Identifier: Japan Registry of Clinical Trials)
Record Dates: First submitted 2024-11-24; First posted 2024-11-27 (Actual); Last update posted 2025-07-02 (Actual); Status verified 2025-07

CONDITIONS: Postherpetic Neuralgia
Keywords: ONO-1110; ONO-1110-04; Postherpetic Neuralgia; PHN
MeSH Terms: conditions — Neuralgia, Postherpetic

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- ONO-1110 (Experimental): ONO-1110 tablets once a day
  Interventions: Drug: ONO-1110
- Placebo (Placebo Comparator): Placebo tablets once daily
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ONO-1110 — ONO-1110 tablets once a day
  Arms: ONO-1110
Drug: Placebo — Placebo tablets once daily
  Arms: Placebo

SUMMARY:
To evaluate the efficacy and safety of ONO-1110 in Japanese patients with postherpetic neuralgia

ELIGIBILITY:
Inclusion Criteria:

* Japanese (both sexes)
* Age (at the time of informed consent): 18 years and older
* Outpatient
* Patients with persistent pain ≥3 months (90 days) after the onset of herpes zoster
* Patients who are considered capable of understanding the study procedures and completing the pain diary and questionnaires appropriately by the investigator (sub-investigator)

Exclusion Criteria:

* Patients who previously underwent neurodestruction or neurosurgical therapy for PHN
* Patients with pain other than PHN that may affect assessments in this study
* Patients with any skin condition related to the site of herpes zoster that may affect assessments in this study
* Patients with a past history of or concurrent neurologic diseases that may affect assessments in this study
* Patients with concurrent psychiatric diseases that may affect assessments in this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2025-02-12 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Change in weekly mean of average pain score (last 7-day mean of past 24-hour average pain scores [NRS] in the pain diary) from baseline to Week 8 of the treatment period | Up to 15 weeks
Adverse Events | Up to 15 weeks

SECONDARY OUTCOMES:
Change in weekly mean of average pain score from baseline to each week | Up to 15 weeks
30%- and 50%-responder rates based on the weekly mean of average pain score (proportions of participants whose weekly mean of average pain score has decreased by 30% and 50% from baseline, respectively) | Up to 15 weeks
Change in weekly mean of worst pain score (last 7-day mean of past 24-hour worst pain scores [NRS] in the pain diary) from baseline to each week | Up to 15 weeks
30%- and 50%-responder rates based on the weekly mean of worst pain score (proportions of participants whose weekly mean of worst pain score has decreased by 30% and 50% from baseline, respectively) | Up to 15 weeks
Change in Brief pain inventory-short form (BPI-SF) score from baseline | Up to 15 weeks
Change in Short Form McGill Pain Questionnaire-2 (SF-MPQ-2) score from baseline | Up to 15 weeks
Patient Global Impression of Change (PGIC) score | Up to 15 weeks
Change in Hospital Anxiety and Depression Scale (HADS) score from baseline | Up to 15 weeks
Plasma ONO-1110 concentrations | Up to 15 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Project Leader, Study Director — Ono Pharmaceutical Co. Ltd
Locations (28):
- Japan (28):
  - Kamezawa Clinic, Aichi
  - Kimura Clinic, Aichi
  - Fukuoka Tokushukai Hospital, Fukuoka
  - Southern Tohoku General Hospital, Fukushima
  - Central Japan International Medical Center, Gifu
  - National Hospital Organization Kure Medical Center, Hiroshima
  - National Hospital Organization Hokkaido Medical Center, Hokkaido
  - Nishinomiya Municipal Central Hospital, Hyōgo
  - Mito Saiseikai General Hospital, Ibaraki
  - Kawasaki Municipal Hospital, Kanagawa
  - Konan Hidamari Pain Clinic, Kanagawa
  - Tai Clinic, Kanagawa
  - Yokohama City Minato Red Cross Hospital, Kanagawa
  - Junwakai Memorial Hospital, Miyazaki
  - Medical Corporation Toyama Dermatology, Miyazaki
  - Yuaikai Tomishiro Chuo Hospital, Okinawa
  - Morimoto Clinic, Osaka
  - Osaka Metropolitan University Hospital, Osaka
  - Medical Corporation Fujigaki Clinic, Ōita
  - Shizuoka Rehabili Pain Clinic, Shizuoka
  - Fukuuchi Pain Clinic, Tokyo
  - Fukuwa Clinic, Tokyo
  - Futaki Skin Care Clinic, Tokyo
  - Juntendo University Hospital, Tokyo
  - Mitaka Pain Clinic, Tokyo
  - Nishiogi Pain Clinic, Tokyo
  - Tokyo-Eki Center-Building Clinic, Tokyo
  - Yamanashi Prefectural Central Hospital, Yamanashi

IPD SHARING:
Plan to Share IPD: No